CLINICAL TRIAL: NCT07407439
Title: A Real-world Study on the Treatment of HR+/HER2- Advanced Breast Cancer Patients With CDK4/6 Inhibitors and Treatment Options After Drug Resistance.
Brief Title: Real-world Studies of CDK4/6 Inhibitors
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJMUCIH-BC-CDK4/6i-01
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Palbociclib; Abemaciclib; Ribociclib; Dalcetrapib; CDK4/6 inhibitors; CDK4/6 inhibitors resistance; HR+/HER2- breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — We will collect the residual tumor samples or peripheral blood samples of the patients in our hospital for genomic and transcriptomic analyses, etc., to prepare for the translational research on the mechanism of CDK4/6i resistance.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Palbociclib cohort: Use palbociclib in combination with endocrine therapy as the treatment regimen.
- Abemaciclib cohort: Use abemaciclib in combination with endocrine therapy as the treatment regimen.
- Ribociclib cohort: Use ribociclib in combination with endocrine therapy as the treatment regimen.
- Dalcetrapib cohort: Use dalcetrapib in combination with endocrine therapy as the treatment regimen.
- Other CDK4/6 inhibitors cohort: Use other CDK4/6 inhibitors in combination with endocrine therapy (including participation in clinical trials of CDK4/6 inhibitors) as the treatment regimen.

SUMMARY:
A single-center, real-world study evaluated the clinical outcomes and safety of CDK4/6 inhibitors combined with endocrine therapy in HR+/HER2- advanced breast cancer, and conducted a summary analysis of the clinical treatment options after the progression of CDK4/6 inhibitors.

DETAILED DESCRIPTION:
This study aims to collect clinical data and case information from real-world clinical practice of patients with HR+/HER2- advanced breast cancer treated with CDK4/6 inhibitors combined with endocrine therapy.

The main research objectives include: 1. To evaluate the differences in efficacy among different CDK4/6 inhibitors combination regimens in advanced patients; 2. To investigate the subsequent treatment options chosen by patients in the real world after progression on CDK4/6 inhibitors, with the aim of constructing a predictive model for the response to subsequent treatments, thereby providing support for clinical decision-making for both doctors and patients in such situations.

The secondary objectives include: 1. To truly reflect the differences in adverse reactions of different CDK4/6 inhibitors in the Chinese population through the collection of laboratory and imaging results; 2. To collect tumor samples or peripheral blood samples from some patients for genomic and transcriptomic analyses, in preparation for translational research on the mechanism of CDK4/6 inhibitors resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Patients diagnosed with HR+/HER2- (as defined by the ASCO/CAP guidelines) advanced breast cancer who were treated in our hospital from March 2022 to March 2025;
3. Received CDK4/6 inhibitors (including but not limited to the four currently marketed ones: palbociclib, abemaciclib, ribociclib, and dalpiciclib) as advanced-stage treatment for at least one cycle;
4. Have complete medical history records, including demographic information, pathological reports, treatment records, laboratory test results, and imaging examination reports, etc.

Exclusion Criteria:

1. Incomplete medical history data.
2. Only received CDK4/6 inhibitors monotherapy.
3. Received CDK4/6 inhibitors as neoadjuvant/postoperative adjuvant intensification therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed as HR+/HER2- (as defined by the ASCO/CAP guidelines) advanced breast cancer between March 2022 to March 2025
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
rwPFS1 and rwPFS2 | 6 weeks
  Real-world progression-free survival (rwPFS1) during treatment with CDK4/6 inhibitors and real-world progression-free survival (rwPFS2) of subsequent treatment lines selected by clinicians after progression on CDK4/6 inhibitor therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Insititute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
At the stage of result publication, we will provide the IPD data in accordance with the specific requirements from the ICMJE journal.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2026-01-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT07407439/Prot_SAP_ICF_000.pdf